CLINICAL TRIAL: NCT00557973
Title: Multiple-Dose Efficacy and Safety Study of XP19986 in Subjects With Spasticity Due to Spinal Cord Injury
Brief Title: A Safety and Efficacy Study of XP19986 in Subjects With Spasticity Due to Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XP-B-065
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Muscle Spasticity
MeSH Terms: conditions — Muscle Spasticity | interventions — BID protein, human; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- XP19986 SR1 10 mg - Placebo (Experimental): Following a 7 day run-in period in which participants take placebo twice a day (BID), participants are randomized to the cohort that will take XP19986 SR1 10 mg BID treatment crossing over to placebo treatment (or the reverse order). Each treatment segment follows the same pattern: 3-9 days of titration, 7 days at target dose, 3-9 days of tapering, followed by a 3-day placebo washout.
  Interventions: Drug: XP19986 SR1, 10 mg BID; Drug: Placebo
- XP19986 SR1 20 mg - Placebo (Experimental): Following a 7 day run-in period in which participants take placebo twice a day (BID), participants are randomized to the cohort that will take XP19986 SR1 20 mg BID treatment crossing over to placebo treatment (or the reverse order). Each treatment segment follows the same pattern: 3-9 days of titration, 7 days at target dose, 3-9 days of tapering, followed by a 3-day placebo washout.
  Interventions: Drug: XP19986 SR1, 20 mg BID; Drug: Placebo
- XP19986 SR1 30 mg - Placebo (Experimental): Following a 7 day run-in period in which participants take placebo twice a day (BID), participants are randomized to the cohort that will take XP19986 SR1 30 mg BID treatment crossing over to placebo treatment (or the reverse order). Each treatment segment follows the same pattern: 3-9 days of titration, 7 days at target dose, 3-9 days of tapering, followed by a 3-day placebo washout.
  Interventions: Drug: XP19986 SR1, 30 mg BID; Drug: Placebo

INTERVENTIONS:
Drug: XP19986 SR1, 10 mg BID — XP19986 Sustained Release (SR) 10 mg tablet dosed orally, twice a day (BID), for approximately 26 days with titration and taper periods
  Other Names: Sustained release Polyox WSR N750, 10 mg
  Arms: XP19986 SR1 10 mg - Placebo
Drug: XP19986 SR1, 20 mg BID — XP19986 Sustained Release (SR) 20 mg tablet dosed orally, twice a day (BID), for approximately 26 days with titration and taper periods
  Other Names: Sustained release Polyox WSR N750, 20 mg
  Arms: XP19986 SR1 20 mg - Placebo
Drug: XP19986 SR1, 30 mg BID — XP19986 Sustained Release (SR) 30 mg tablet dosed orally, twice a day (BID), for approximately 26 days with titration and taper periods
  Other Names: Sustained release Polyox WSR N750, 30 mg
  Arms: XP19986 SR1 30 mg - Placebo
Drug: Placebo — Placebo tablets to match active intervention, taken twice a day (BID) for approximately 26 days with titration and taper periods. Also taken during placebo washout periods.
  Other Names: sugar pill

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of treatment with XP19986 Sustained Release (SR) Tablet compared to placebo in subjects with spasticity due to spinal cord injury

DETAILED DESCRIPTION:
This is a multiple-dose, randomized, placebo-controlled crossover study of the efficacy and safety of XP19986 SR1 in subjects with spasticity due to spinal cord injury. Three cohorts of subjects are randomized to receive XP19986 SR1 10 mg every 12 hrs or 20 mg every 12 hrs or 30 mg every 12 hrs in one treatment segment and placebo every 12 hrs in the alternate treatment segment. Each subject serves as their own control in this cross-over study.

ELIGIBILITY:
Inclusion Criteria:

* Spasticity secondary to traumatic spinal cord injury between C-5 and T-12 spinal cord levels, at least 12 months post-injury with a stable neurological deficit

Exclusion Criteria:

* Traumatic brain injury or cognitive deficit of any etiology that may influence compliance with study procedures or outcome measures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Maximum Ashworth score | Day 17
  Ashworth score for each treatment segment before dosing and 2, 4, and 6 hours after the morning dose. Evaluate the difference in the primary endpoint between active and placebo treament segments at 17th day of dosing in each segment

SECONDARY OUTCOMES:
Average Ashworth score | Day 17
  This was the average of Ashworth scores obtained on Day 17 of dosing across 6 muscle groups for each treatment segment before dosing and 2, 4, and 6 hours after the morning dose
Two Highest Ashworth scores | Day 17
  This was the average of Ashworth scores obtained on Day 17 of dosing from the muscle groups that had the 2 highest Ashworth scores at baseline for each treatment segment before dosing and 2, 4, and 6 hours after the morning dose
Average Non-zero Ashworth Scores | Day 17
  This was the average of Ashworth scores obtained on Day 17 of dosing from the muscle groups that had a non-zero Ashworth score at baseline for each treatment segment before dosing and 2, 4, and 6 hours after the morning dose

CONTACTS AND LOCATIONS:
Overall Officials: Michael Leong, M.D., Study Director — XenoPort, Inc.
Locations (11):
- United States (11):
  - Downey, California
  - Gilroy, California
  - Pasadena, California
  - San Jose, California
  - Englewood, Colorado
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - Ann Arbor, Michigan
  - Detroit, Michigan